CLINICAL TRIAL: NCT00429286
Title: Preserving Function in Rural Breast Cancer Patients Undergoing Chemotherapy
Brief Title: Preserving Function in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 1R03CA124200-01 (NIH)
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Breast Cancer
Keywords: Health Services Research
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Problem Solving Training — A systematic cognitive-behavioral intervention teaching problem solving skills for addressing functional impairment related to breast cancer and its treatment.

SUMMARY:
Breast cancer patients experience functional limitations related to the cancer and treatment side effects. Early functional limitations affect short- and long-term quality of life, and may lead to long-term complications. Patients living in rural areas are at particular risk because they do not have easy access to services. Therefore, early intervention is indicated to have an impact on the overall public health. Problem solving training (PST) is a standardized manual driven intervention that may be ideally suited to assist breast cancer patients to preserve their valued activities and to comply with recommended symptom management regimens (e.g., physical therapy, aerobic exercise and relaxation/guided imagery) that improve function. Telephone-based PST provided from a centralized location (such as the comprehensive cancer center) may improve access and outcomes in a cost-effective manner. We propose to conduct a feasibility study of a PST intervention with 30 rural breast cancer patients undergoing adjuvant treatment randomly assigned to PST or to usual care. The intervention group will receive weekly phone-based PST sessions for six consecutive weeks. The specific aims of this R03 small grant application are to:1) Test the feasibility of enrolling and retaining newly diagnosed breast cancer patients in a clinical trial to assess telephone-based PST. 2) Collect preliminary data on outcome measures of function to determine effect size estimates that will inform power analyses for a full scale randomized controlled study. Primary outcome measures will be acceptance rates for enrollment in the study, retention rates across both intervention arms, and satisfaction levels with the PST intervention. Assessments will be conducted at baseline, and at six weeks (end of PST intervention) and 3 months following baseline. The long-term goal of this line of investigation is to develop practical, widely applicable rehabilitation models of care to preserve function and decrease distress in cancer patients undergoing treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Females, age > 18 years.
2. First breast cancer diagnosis, Stages 1-3.
3. Beginning the second chemotherapy cycle.
4. English speaking and literate.

Exclusion Criteria:

1. Previous or concurrent malignancy, except for non-melanotic skin cancers.
2. Lifetime diagnosis of schizophrenia or bipolar disorder.
3. Moderate-severe cognitive impairment indicated by a score < 3 on a 6-item cognitive screener.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients undergoing chemotherapy at the Norris Cotton Cancer Center in Lebanon, NH.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark T Hegel, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States